CLINICAL TRIAL: NCT03725553
Title: A Randomized Clinical Trial Examines the Efficacy of Intra-myometrial Local Injection of Vasopressin to Reduces the Blood Loss During Cesarean Section in Placenta Previa
Brief Title: Intra-myometrial Vasopressin During Cesarean Section in Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu 192/7/18
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Placenta Previa
Keywords: vasopressin; placenta previa; postpartum hemorrhage
MeSH Terms: conditions — Placenta Previa; Diabetes Insipidus; Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients were randomized to two groups, patients according to a two -blocked randomization list which was coded (1 or 2) at 1:1 ratio. The study drug was administered immediately after delivery, as soon as the umbilical cord was clamped. The experimental group received a bolus injection of vasopressin (4 IU) diluted to 2 mL with saline into the myometrium of the placental bed during slow (30-s) Conversely, the placebo group received a 10-mL bolus injection of saline into the myometrium during slow (30-seconds).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramyometrial Vasopressin (Experimental): the experimental group received a bolus injection of vasopressin (4 IU) diluted to 2 mL with saline into the myometrium of the placental bed during slow (30-seconds) immediately after delivery, as soon as the umbilical cord was clamped.
  Interventions: Drug: Intramyometrial Vasopressin
- Placebo (Placebo Comparator): the placebo group received a 10-mL bolus injection of saline into the myometrium during slow (30-seconds)immediately after delivery, as soon as the umbilical cord was clamped.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intramyometrial Vasopressin — a bolus injection of vasopressin (4 IU) diluted to 2 mL with saline into the myometrium of the placental bed during slow (30-seconds) immediately after delivery, as soon as the umbilical cord was clamped.
  Other Names: Experimental
  Arms: Intramyometrial Vasopressin
Drug: Placebo — the group received a 10-mL bolus injection of saline into the myometrium during slow (30-seconds)as soon as the umbilical cord was clamped.
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
Placenta previa can have serious adverse consequences for the mother, including an increased risk of maternal mobility, antenatal and intrapartum hemorrhage, and the mother may, therefore, require a blood transfusion or even an emergency hysterectomy. Although it is a relatively rare condition with an overall incidence of 0.28-2.0% of all deliveries, it has been suggested that the incidence of placenta previa is increasing. Many gynecological surgeons use a local injection of vasopressin, which is a known peripheral vasoconstrictor, at the time of laparoscopic myomectomy to decrease blood loss. In addition, the useful role for local infiltration of vasopressin to arrest hemorrhage from the placental bed has been demonstrated in several obstetrical case reports. The vasopressin V1α receptor has been demonstrated to be present in the myometrium of both non-pregnant and pregnant women and contributes to myometrial contraction. Therefore, the investigators evaluated the effect of local injection of vasopressin on the blood loss and secondary impact on complications during cesarean section in cases of placenta previa.

DETAILED DESCRIPTION:
The study drug was administered immediately after delivery, as soon as the umbilical cord was clamped. The experimental group received a bolus injection of vasopressin (4 IU) diluted to 2 mL with saline into the myometrium of the placental bed during slow (30-seeconds) Conversely, the placebo group received a 10-mL bolus injection of saline into the myometrium during slow (30-seconds).

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a single term fetus scheduled for an elective cesarean section for complete placenta previa and invited them to participate in the study. The placenta previa was defined as a placenta completely covering the cervical os in ultrasound examination

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease.
* patients with the high possibility of the morbid adherent placenta.
* known coagulopathy
* those presented with severe antepartum hemorrhage will be excluded
* hypersensitivity or contraindications of use of vasopressin
* patient refuses to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant patients scheduled for cesarean section for placenta previa
Enrollment: 120 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 6 hours post operative
  blood loss > 1000ml measured by direct and gravimetric methods

SECONDARY OUTCOMES:
intraoperative blood loss | during the operation
  amount of blood loss during cesarean section
The number of participant needed for blood transfusion | 24 hours post operative
  Calculation of the number of participant needed for blood transfusion
need of extra surgical maneuvers | during the operation
  internal iliac ligation or hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No